CLINICAL TRIAL: NCT01793272
Title: Beneficial Effect of Adding Pentoxifylline to Processed Semen Samples on ICSI Outcome in Infertile Males With Mild and Moderate Asthenozoospermia: Randomized Controlled Prospective Crossover Study
Brief Title: Beneficial Effect of Adding Pentoxifylline to Processed Semen Samples on ICSI Outcome in Infertile Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adam International Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Raef Sadek, Ahmad Raef, Adam International Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-2-13
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Pentoxifylline Allergy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pentoxifylline (Other): effect of pentoxifylline on ICSI outcome
  Interventions: Other: effect of pentoxifylline on ICSI outcome

INTERVENTIONS:
Other: effect of pentoxifylline on ICSI outcome — semen processing with pentoxifylline prior to ICSI

SUMMARY:
To evaluate the effect of pentoxifylline used in preparation of semen samples that will be used for ICSI in infertile men complaining of mild and moderate asthenozoospermia (i.e. cases which does not need motility enhancement prior to ICSI) in comparison to semen samples without pentoxifylline preparation on the outcome of ICSI.

DETAILED DESCRIPTION:
The primary outcome measures were the number of oocytes retrieved, the number of oocytes injected, number of oocytes fertilized, fertilization rate, number of embryos and their quality (G1: good embryos, G2: fair embryos and G3: bad embryos), number of embryos transferred (ET), number of embryo sacs, embryo implantation rate, pregnancy rate and abortion rate for all 3 groups and pregnancy rate and abortion rate for both group (I) and group (II).

ELIGIBILITY:
Inclusion Criteria:

* seeking ICSI for infertility

Exclusion Criteria:

* Pyospermia, presence of antisperm antibodies. Azoospermia, severe male factor, severe asthenozoospermia. Past history of orchitis. Patients who received empirical treatment for asthenozoospermia e.g. oral Pentoxifylline, l-carnitine or antioxidants during the past 3 to 6 month. Diabetics, hypertensives or patients with any other chronic systemic illnesses. Wife's age more than 35 years. Low antral count. Presence of any ovarian factor contributing to infertility e.g. polycystic ovaries.

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
ICSI outcome | from October 2010 to April 2011.

CONTACTS AND LOCATIONS:
Overall Officials: Medhat Amer, MD, Study Director — M.Amer
Locations (1):
- Adam International Hospital, Giza, Giza Governorate, Egypt

REFERENCES:
- [Derived] Amer M, Metawae B, Hosny H, Raef A. Beneficial effect of adding pentoxifylline to processed semen samples on ICSI outcome in infertile males with mild and moderate asthenozoospermia: A randomized controlled prospective crossover study. Iran J Reprod Med. 2013 Nov;11(11):939-44. PMID 24639720